CLINICAL TRIAL: NCT00095654
Title: The DREAM (Diabetes Reduction Assessment With Ramipril and Rosiglitazone Medication) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gerstein, Hertzel, MD (Individual)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Aventis Pharmaceuticals (Industry); GlaxoSmithKline (Industry); King Pharmaceuticals is now a wholly owned subsidiary of Pfizer (Industry); Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: DREAM30Nov2002
Record Dates: First submitted 2004-11-05; First posted 2004-11-08 (Estimated); Last update posted 2009-11-10 (Estimated); Status verified 2009-11

CONDITIONS: Impaired Glucose Tolerance; Cardiovascular Disease; Glucose Metabolism Disorders
Keywords: diabetes prevention; ramipril; rosiglitazone; impaired glucose tolerance; isolated impaired fasting glucose; Isolated Impaired Glucose Tolerance
MeSH Terms: conditions — Glucose Intolerance; Cardiovascular Diseases; Glucose Metabolism Disorders | interventions — Ramipril; Rosiglitazone

INTERVENTIONS:
Drug: Ramipril
Drug: Rosiglitazone

SUMMARY:
The purpose of this study is to determine if ramipril and/or rosiglitazone prevent the onset of type 2 diabetes.

DETAILED DESCRIPTION:
The DREAM trial is a large, international, multi-centre, randomized double-blind controlled trial. A total of at least 4000 participants with impaired glucose tolerance (IGT) and 1000 participants with isolated impaired fasting glucose (IIFG) will be recruited from major international centres over an 18 month period. They will be randomly allocated to either ramipril and/or rosiglitazone using a 2X2 factorial design and followed for at least 3 years after randomization. Participants will be assessed at regular intervals to ascertain the occurrence of the primary outcome (new onset diabetes mellitus or all cause mortality) and other secondary outcomes. A diagnosis of diabetes will be made if 2 consecutive plasma glucose levels exceed the diagnostic thresholds (i.e. a fasting plasma glucose >=7.0 mmol/l (126 mg/dl) or a 2 hr plasma glucose >=11.1 mmol/l (200 mg/dl)) within a 3 month period. Assuming an annual event rate of 5%, this sample size provides 90% power to detect a 22% reduction in the rate of the primary outcome.

Potential Significance of the Study: This study could provide new strategies for the prevention of type 2 diabetes as well as provide insight into the relationship between cardiovascular disease and diabetes.

Study Update: A total of 5269 participants were enrolled into the study. 4527 Participants had IGT and 739 participants had IIFG. The study is currently in the follow-up phase.

DREAM On

In order to determine whether or not the benefits observed during the active phase of the trial are sustained after cessation of active medication use, further follow-up of the DREAM cohort will be conducted in the passive DREAM ObservatioN (DREAM On) follow-up study.

DREAM On will assess approximately 1500 consenting DREAM participants without a diagnosis of diabetes at the end of the washout phase after a post-trial period of between 1 and 2 years to determine the effect of on-trial exposure to rosiglitazone and/or exposure to ramipril on: a) the primary outcome (incident diabetes or death); and b) regression or maintenance of normoglycemia. Participants will be free to take any medications that are indicated and may participate in other research studies, according to the judgment of their own physician.

ELIGIBILITY:
Inclusion Criteria:

* impaired glucose tolerance (FPG < 7 mmol/L or 126 mg/dL AND 2 hr PG >= 7.8 mmol/L and < 11.1 mmol/L (140 mg/dL and < 200 mg/dL)or,
* isolated impaired fasting glucose (FPG >= 6.1 mmol/L and < 7 mmol/L (FPG >= 95 mg/dL and < 126 mg/dL) AND 2 hr PG < 7.8 mmol/L (140 mg/dL).

Exclusion Criteria:

* current use of an ACE-inhibitor (ACE-I) or thiazolidinedione(TZD)
* known hypersensitivity to ACE-I
* prior use of anti-diabetic medications (with the exception of during pregnancy)
* use of systemic glucocorticoids or niacin
* congestive heart failure or EF < 40%
* existing cardiovascular disease (previous MI, stroke, angina, uncontrolled hypertension)
* diabetes
* renal or hepatic disease
* major illness
* use of another experimental drug
* pregnant or unwilling to use reliable contraception
* major psychiatric disorder
* diseases that affect glucose tolerance
* unwillingness to be randomized or sign informed consent
* known uncontrolled substance abuse
* inability to communicate with research staff

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5000
Dates: Start 2001-07; Study Completion 2006-10 (Actual)

PRIMARY OUTCOMES:
diabetes
death

SECONDARY OUTCOMES:
Myocardial infarction (MI)
Stroke
Congestive Heart Failure
Angina
Revascularization procedures
Ventricular Arrhythmia
Renal Events

CONTACTS AND LOCATIONS:
Overall Officials: Salim Yusuf, MD, Principal Investigator — McMaster University, FAX # 905-521-1166; Hertzel Gerstein, MD, Principal Investigator — McMaster University, FAX # 905-521-4967

REFERENCES:
- [Background] Gerstein HC, Yusuf S, Holman R, Bosch J, Pogue J; DREAM Trial Investigators. Rationale, design and recruitment characteristics of a large, simple international trial of diabetes prevention: the DREAM trial. Diabetologia. 2004 Sep;47(9):1519-27. doi: 10.1007/s00125-004-1485-5. Epub 2004 Aug 21. PMID 15322749
- [Result] DREAM Trial Investigators; Bosch J, Yusuf S, Gerstein HC, Pogue J, Sheridan P, Dagenais G, Diaz R, Avezum A, Lanas F, Probstfield J, Fodor G, Holman RR. Effect of ramipril on the incidence of diabetes. N Engl J Med. 2006 Oct 12;355(15):1551-62. doi: 10.1056/NEJMoa065061. Epub 2006 Sep 15. PMID 16980380
- [Result] DREAM (Diabetes REduction Assessment with ramipril and rosiglitazone Medication) Trial Investigators; Gerstein HC, Yusuf S, Bosch J, Pogue J, Sheridan P, Dinccag N, Hanefeld M, Hoogwerf B, Laakso M, Mohan V, Shaw J, Zinman B, Holman RR. Effect of rosiglitazone on the frequency of diabetes in patients with impaired glucose tolerance or impaired fasting glucose: a randomised controlled trial. Lancet. 2006 Sep 23;368(9541):1096-105. doi: 10.1016/S0140-6736(06)69420-8. PMID 16997664
- [Derived] Natale P, Palmer SC, Navaneethan SD, Craig JC, Strippoli GF. Angiotensin-converting-enzyme inhibitors and angiotensin receptor blockers for preventing the progression of diabetic kidney disease. Cochrane Database Syst Rev. 2024 Apr 29;4(4):CD006257. doi: 10.1002/14651858.CD006257.pub2. PMID 38682786
- [Derived] DREAM Trial Investigators. Incidence of diabetes following ramipril or rosiglitazone withdrawal. Diabetes Care. 2011 Jun;34(6):1265-9. doi: 10.2337/dc10-1567. Epub 2011 Apr 22. PMID 21515846
- [Derived] DREAM Trial Investigators; Dagenais GR, Gerstein HC, Holman R, Budaj A, Escalante A, Hedner T, Keltai M, Lonn E, McFarlane S, McQueen M, Teo K, Sheridan P, Bosch J, Pogue J, Yusuf S. Effects of ramipril and rosiglitazone on cardiovascular and renal outcomes in people with impaired glucose tolerance or impaired fasting glucose: results of the Diabetes REduction Assessment with ramipril and rosiglitazone Medication (DREAM) trial. Diabetes Care. 2008 May;31(5):1007-14. doi: 10.2337/dc07-1868. Epub 2008 Feb 11. PMID 18268075